CLINICAL TRIAL: NCT03983798
Title: Learning Process of 5th Year Medical Students During Simulation Training in Psychiatry: a Multicentric Mixed Method Study
Brief Title: Learning Process of Medical Students During Simulation Training in Psychiatry
Acronym: APSIMP
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: PSY-04-2018
Record Dates: First submitted 2018-10-16; First posted 2019-06-12 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-07

CONDITIONS: Role Playing; Psychology; Learning
Keywords: Simulation training; Patient simulation; Psychiatric; Medical students; Educational; Medical
MeSH Terms: interventions — Psychiatry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Simulation training in psychiatry: Convenient sample of 72 voluntary medical students, allocated among 6 groups of around 12 students, will be recruited at Paris Descartes, Paris Diderot and Brest Universities between september of 2018 and June of 2019.
  Interventions: Other: Simulation training in psychiatry

INTERVENTIONS:
Other: Simulation training in psychiatry — Each participant will complete 6 hours of psychiatric simulation training, dealing with mood disorders, anxious disorders, eating disorders, borderline disorders, substance abuse and schizophrenia. Simulation training will be supplemented by brief lecture on concept map and portfolio at the beginning of the first hour.
  Curriculum integration of simulation training in psychiatric course assure that each pathology studied is supplemented by a one-hour lecture and 1 to 3 hours clinical cases and MCQ training. A part of the medical students are supplemented by clinical practice ; whereas the other won't benefit from clinical practice.

SUMMARY:
In french context, simulation training is not well implemented in medical school, mainly in psychiatry. We aim to build a formative and summative assessment tool of competences specific to this pedagogic context, so as to support its development.

This studies aims to explore learning process and factors supporting or preventing from learning of medical students during simulation in psychiatry.

A convenient sample of 72 voluntary participants, allocated among 6 groups of around 12 students, will be recruited at Paris Descartes, Paris Diderot and Brest Universities between september of 2018 and june of 2019. Each participant will complete 6 hours of psychiatric simulation training, dealing with mood disorders, anxious disorders, eating disorders, borderline disorders, substance abuse and schizophrenia.

Participant will be offered to complete a portfolio about learning process during the trimester they are involved, a concept gap before and after each training and the " Learning Effectiveness Inventory Scale "at the end of simulation. A purposive sample of students will have to complete a face-to-face semi-interview (until reaching data saturation).

Video record of simulation and audio-record of debriefing will be analysed to enhance triangulation process of analysis.

DETAILED DESCRIPTION:
Since the end of the nineties, pedagogical transformations question traditional pedagogical system which supports a passive learning from master to student, trying to overcome classical " teaching paradigm" to " learning paradigm ". Despite several critics, the notion of " professional competence " emerges as one of the essential purpose of learning. Competence might be defined as " complex ability that professional built, starting from a specialized knowledge base, developed and controlled by a collegial peer who constitute the profession ", implying " a reflexive practice inside and after action " which creates or increases new competence in return.

However in french context, this paradigmatic revolution didn't really happened yet, including in psychiatry. Moreover, there are no engineering didactic work on specific skills required by a physician (psychiatrist or not) should have in care of a patient with psychiatric disorders. For instance, skills required when a surgeon has to deliver a "clear, loyal and adjusted" information to a patient with a schizophrenia ; and try to get his or her agreement so as to operate a intestinal blockage? As a matter of facts, no integrated competence referential will be able to be a reference in this work.

In a report which is nowadays a reference for the faculties of medicine all over the world, the Royal College of Physicians and Surgeons of Canada (CRMCC) define a framework of essential skills that each physician have to control: medical expertise, erudition ; communicational and relational abilities; collaboration ; professionalism ; management; health promotion. In the French context, skills that each medical student have to provide fo the psychiatric speciality are defined by 33 questions of national classifying exam (ECN). The " Psychiatry and Addictology Referential " points to medical students the reference knowledge to provide to respond to these questions during the challenge of ECN. But this referential doesn't explain skills, abilities and attitudes required with a patient with psychiatric disorders.

The places of providing essential skills defined by CRMCC applied in French psychiatry (as relational and communicational skills for instance) are thus often situated in others spaces. Realization of well supervised clerkship in psychiatry constitutes for example one of the privilege way of skills acquisition. Nonetheless in French context, all the undergraduate students can benefit from psychiatry during their clerkship; especially because of the rarefaction of well supervised internship (decreasing demography of psychiatrist), associated with increase number of medical student over the past few years. Moreover, realization of an only internship can not include all the diversity of main family situation that should be known by each physician; mainly because of dichotomy of internship between adult and child and adolescent psychiatry, specific populations specific who go to different service according to there trouble (emergencies, closed unit, expert diagnosis centers…). Providing pedagogical tools allowing acquisition of basic skills, abilities and attitudes (complementary to knowledge and know-repeat) to care patient with psychiatric disorders seems thus interesting, for improving medical training.

Besides, assessment modalities determine for students work methodology and time involved in each learning, following Hawthorne effect. Assessments support learning assessed, involving long term memory, following " testing effect " ; and hierarchize planning of ulterior learning activities. Trials of ECN in this current shape will probably value acquisition of declarative knowledge for students who would like to succeed in the competition; to the detriment of know-how and life skills. These skills to care patients who suffer from psychiatric disorders won't be neither provided during a specialty residency, unless it might be especially oriented to psychiatry. Thus, it seems important to wider summative assessment modalities in psychiatry during undergraduate medical studies, so as to value acquisition of the wall skills required for a physician in care of a patient with psychiatric disorders. Which implies precise explanation of skills, abilities and attitudes needed, to balance success of ECN with their acquisition. In that context, simulation can offer a good response to this double aim : formative et summative. However, if some theorical approach are references to understand learning process in simulation, very few learning tool are validated in simulation, and none, to our knowledge, did a modelisation on learning process in psychiatric simulation for medical students.

Objectives:

This study aims to explore learning process in a simulation training using simulated patients in psychiatry for 5th year medical students.

This study is one of the 3 studies included in a PhD on learning process during simulation training in psychiatry.

The results of this 3 studies will aim at building a formative and summative assessment tool of competences specific to this pedagogic context

Methodology:

A convenient sample of 72 voluntary medical students, allocated among 6 groups of around 12 students, will be recruited at Paris Descartes, Paris Diderot and Brest Universities between september of 2018 and june of 2019. Each participant will be offered to complete 6 hours of psychiatric simulation training, dealing with mood disorders, anxious disorders, eating disorders, borderline disorders, substance abuse and schizophrenia.

Study design is a mixted method study, following grounded theory including:

* Quantitative features:

  * Pre/post test concept map
  * Self-reported questionnaires : " Learning Effectiveness Inventory Scale "
  * Sociodemographical data and others questions
* Qualitative : Grounded Theory

  * Semi-structured interview of learners
  * Portfolio completed during clinical clerkship, after simulation on each pathology studied
  * Pre/post test concept map (for clinical reasonning features)
  * Video-record of simulation
  * Audio-record of briefing and debriefing

ELIGIBILITY:
Inclusion Criteria:

* Age > to 18 years old
* Undergraduate medical student of Paris Descartes, Paris Diderot or Brest University
* During university year 2018-2019
* French or English langage
* Agreement

Exclusion Criteria:

•Refusal of agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Voluntary medical students recruited at Paris Descartes, Paris Diderot and Brest Universities
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Learning process assessed by qualitative approach ( constructivist Grounded Theory) through semi-structured interviews. | 6 weeks
  Learning process assessed by semi-structured face-to-face interview from a purposive sample of participants, until reaching data saturation. There are no scale, no score, we have just to follow this qualitative method of analysis (Glaser BG, Strauss AL. The discovery of grounded theory: Strategies for qualitative research. Chicago: Aldine; 1967).
Learning process assessed by qualitative approach ( constructivist Grounded Theory) through written port-folio. | 6 weeks
  Learning process assessed on written port-folio with open questions on learning process on each simulation session, until reaching data saturation.There are no scale, no score, we have just to follow this qualitative method of analysis (Glaser BG, Strauss AL. The discovery of grounded theory: Strategies for qualitative research. Chicago: Aldine; 1967).

SECONDARY OUTCOMES:
Factors supporting or preventing learning of 5th year medical students during simulation training in psychiatry assessed by qualitative approach ( constructivist Grounded Theory) through semi-structured interviews. | 6 weeks
  Factors supporting or preventing learning process assessed by semi-structured face-to-face interview from a purposive sample of participants, until reaching data saturation.There are no scale, no score, we have just to follow this qualitative method of analysis (Glaser BG, Strauss AL. The discovery of grounded theory: Strategies for qualitative research. Chicago: Aldine; 1967).
Factors supporting or preventing learning of 5th year medical students during simulation training in psychiatry assessed by qualitative approach ( constructivist Grounded Theory) through written port-folio. | 6 weeks
  Factors supporting or preventing learning process assessed on written port-folio with open questions on factors supporting or preventing from learning process on each simulation , until reaching data saturation.There are no scale, no score, we have just to follow this qualitative method of analysis (Glaser BG, Strauss AL. The discovery of grounded theory: Strategies for qualitative research. Chicago: Aldine; 1967).
Evolution of concept map on main psychiatric disorders studied during psychiatric simulation. | Before and immediately after simulation
  Quantitative and qualitative analysis of concept map to understand cognitive reasoning.There are no consensual and validated method to assess cognitiv reasoning with concept map for the time being. There is 3 method tried to assess mind map. We plan to compute these method with qualitative approach.
Satisfaction about learning: Self-questionnaire | Immediately after the end of simulation
  Self-questionnaire: "Simulation Learning Effectiveness Inventory" (SLEI), divided in 7 different section with 32 questions. Each question is quoted on a 5-points Lickert scale (1 for not at all; 5 for "totaly agree"). Results are reported individually for each question, or by a mean on 5-points Lickert scale for each section: course; ressource; debrief; clinical ability; confidence; problem solving; collaboration.
  (Chen SL, Huang TW, Liao I-c, Liu C. Development and validation of the Simulation Learning Effectiveness Inventory. Journal of advanced nursing. 2015;71(10):2444-53.)
Sociodemographic and other questions | Immediately after the end of simulation
  Age, gender, previous experience in simulation, in psychiatry and in psychiatric simulation, first, second and third specialty choice

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Aude PIOT, MD, PhD, Principal Investigator — Institut Mutualiste Montsouris
Locations (2):
- France (2):
  - Institut mutualiste montsouris, Paris
  - Institut Mutualiste Montsouris, Paris, Île-de-France Region

REFERENCES:
- [Background] Lavoie P, Michaud C, Belisle M, Boyer L, Gosselin E, Grondin M, Larue C, Lavoie S, Pepin J. Learning theories and tools for the assessment of core nursing competencies in simulation: A theoretical review. J Adv Nurs. 2018 Feb;74(2):239-250. doi: 10.1111/jan.13416. Epub 2017 Sep 20. PMID 28815750
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Chen SL, Huang TW, Liao IC, Liu C. Development and validation of the Simulation Learning Effectiveness Inventory. J Adv Nurs. 2015 Oct;71(10):2444-53. doi: 10.1111/jan.12707. Epub 2015 Jun 15. PMID 26073864